CLINICAL TRIAL: NCT02251184
Title: Comparison of Pharmacokinetics of Dipyridamole Administered as Aggrenox® (Dipyridamole Extended Release Plus Aspirin) Capsule Versus Dipyridamole Immediate Release Plus Aspirin Following Alteration of Stomach pH by the Prior Administration of a Proton-pump Inhibitor: An Open-label 2-way Randomized Cross-over Study in Healthy Male and Female Subjects Age 40-65.
Brief Title: Pharmacokinetics of Dipyridamole Administered as Aggrenox® (Dipyridamole Extended Release Plus Aspirin) Capsule Versus Dipyridamole Immediate Release Plus Aspirin Following Alteration of Stomach pH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9.146
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — Aspirin, Dipyridamole Drug Combination; Dipyridamole; Aspirin; Lansoprazole

ARMS (2):
- Aggrenox (Experimental): extended release
  Interventions: Drug: Aggrenox; Drug: Lansoprazole
- dipyridamole+aspirin (Active Comparator): immediate release
  Interventions: Drug: Dipyridamole; Drug: Aspirin; Drug: Lansoprazole

INTERVENTIONS:
Drug: Aggrenox
  Arms: Aggrenox
Drug: Dipyridamole
  Arms: dipyridamole+aspirin
Drug: Aspirin
  Arms: dipyridamole+aspirin
Drug: Lansoprazole

SUMMARY:
Comparison of pharmacokinetics of dipyridamole administered as Aggrenox versus dipyridamole administered as the immediate release formulation plus aspirin, under conditions of reduced stomach acidity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age 40 - 65 years, inclusive, at time of Visit 1
* Stomach pH > 4.0 on three consecutive measurements separated by at least five minutes, measured at Visits 3B and 5B prior to dosing with Aggrenox or dipyridamole-aspirin (DP-ASA)

Exclusion Criteria:

* Any findings of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and considered by the investigator to be of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders considered by the investigator to be of clinical relevance
* History of gastro-intestinal ulcer, perforation or bleeding
* Surgery of the gastro-intestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy), neurological disorders, or psychiatric disorders
* Chronic or relevant acute infections. Screening tests will be performed for HIV, hepatitis B, and hepatitis C
* History of hypersensitivity to Aggrenox or any of the components or excipients
* Intake of drugs with a long dominant half-life (>24 hours) 1 month or less prior to Visit 1
* Use of any drugs which might influence the results of the trial ten days or less prior to Visit 1
* Participation in another trial with an investigational drug 1 month or less prior to Visit 1
* Known alcohol abuse
* Known drug abuse (a drug screening test will be performed at Visits 1, 3, and 5)
* Blood donation 1 month or less prior to Visit 1
* Excessive physical activities five days or less prior to Visit 1
* History of hemorrhagic diathesis
* History of bronchial asthma
* Any laboratory value outside the reference range, considered by the investigator to be of clinical relevance

For female subjects:

* Nursing
* Pregnancy
* Positive pregnancy test
* No adequate contraception (adequate contraception includes sterilization, intrauterine device, or oral contraceptives)
* Inability to maintain adequate contraception during the whole study period

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2000-10; Primary Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
area under the concentration time curve (AUC0-12) | up to 12 hours

SECONDARY OUTCOMES:
area under the concentration time curve 0-48 hours (AUC0-48) | up to 48 hours
area under the concentration time curve extrapolated to infinity (AUC0-inf) | up to 3 days
maximum observed plasma concentration (Cmax) | up to 3 days
time to maximum observed plasma concentration (Tmax) | up to 3 days
terminal half life (t1/2) | up to 3 days
number of subjects with adverse events | up to 3 weeks
number of subjects with clinically significant changes in laboratory findings | up to 17 days